CLINICAL TRIAL: NCT00766909
Title: Diabetogenicity of Cyclosporine and Tacrolimus
Acronym: CSATAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: M-20080060
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Complications of Transplanted Organs and Tissue; Diabetes Mellitus Nos New Onset
Keywords: Insulin pulsatility; Insulin secretion; Insulin sensitivity; Calcineurin inhibitor; Cyclosporine; Tacrolimus
MeSH Terms: conditions — Insulin Resistance | interventions — Cyclosporine; Tacrolimus; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CsA (Experimental): Cyclosporine
  Interventions: Drug: cyclosporine
- Tac (Experimental): Tacrolimus
  Interventions: Drug: tacrolimus
- Placebo (Placebo Comparator): placebo/saline
  Interventions: Other: Capsules and isotonic saline

INTERVENTIONS:
Drug: cyclosporine — For Healthy volunteers (study 1) and Dialysis patients (study 2): Single intravenous infusion of 0.155 mg/kg over a maximum duration of 5 hours.
  For Dialysis Patients (study 2): Oral intake of 4 mg/kg 2 times daily for 8-11 days.
  Other Names: Sandimmun
  Arms: CsA
Drug: tacrolimus — For Healthy volunteers (study 1) and Dialysis patients (study 2): Single intravenous infusion of 0.0012 mg/kg over a maximum duration of 5 hours.
  For Dialysis Patients (study 2): Oral intake of 0.1 mg/kg 2 times daily for 8-11 days.
  Other Names: Prograf
  Arms: Tac
Other: Capsules and isotonic saline — For Healthy volunteers (study 1) and Dialysis patients (study 2): Single intravenous infusion of 0.06 ml/kg isotonic saline over a maximum duration of 5 hours.
  For Dialysis patients (study 2): Placebo capsules 2 times daily for 8-11 days.
  Other Names: Saline; NaCl
  Arms: Placebo

SUMMARY:
Cyclosporine (CsA) and Tacrolimus (Tac) are immunosuppressive agents comprising the cornerstone of treatment among organ transplant recipients. Unfortunately diabetes is a known complication after transplantation, yet the underlying mechanisms of this type of diabetes are still unresolved. A direct comparison of the diabetogenic effects of CsA and Tac, without interference of corticosteroid treatment, has not yet been investigated using a hyperinsulinemic euglycemic glucose clamp technique, which is the best method for estimating insulin sensitivity.

Randomized, investigator-blinded cross-over studies will be carried out, studying 10 healthy subjects and 10 hemodialysis patients. Each participant will receive treatment with CsA, Tac and placebo respectively in a random order. The results will be of relevance to the choice and monitoring of immunosuppressive regimens in kidney transplant recipients as well as the development of better treatment modalities for diabetes.

DETAILED DESCRIPTION:
Background: Post-transplantation diabetes mellitus (PTDM) is a complication of the calcineurin inhibitors (CI) cyclosporine (CsA) and Tacrolimus (Tac), but much controversy still exists regarding the mechanism leading to this disorder. Several studies using intravenous (IVGTT) or oral glucose tolerance tests have shown that CsA and Tac tend to reduce insulin release, while corticosteroids increase insulin resistance. Decreased insulin secretion may be the result of beta-cell toxicity, apoptosis or inhibition of calcineurin signaling cessating insulin gene transcription. Comparing the drug using IVGTT has shown that long-term glucose metabolism is not significantly different between the two. Reviewing the literature brings forth that some of these data and the observed higher incidence of PTDM in Tac-treated recipients are conflicting.

To or knowledge, comparison of the diabetogenic effects of CsA and Tac, without concomitant corticosteroids, has never been investigated using the gold standard to estimate insulin sensitivity; a hyperinsulinemic euglycemic glucose clamp (HEGC).

Hypotheses: CsA and Tac are able to induce diabetes, by exerting acute and chronic effects on pancreas beta-cell performance and insulin sensitivity.

The hypothesized effects will be investigated during following studies:

1. Acute effect in 10 healthy subjects undergoing HEGC
2. Chronic effect in 10 pre-transplant uremic patients undergoing HEGC

Methods: The studies are randomized, double-blinded (Study 1) and investigator blinded (Study 2) cross-over designs. Each study subject participates in three experimental study days with an interval of 4-6 weeks. A HEGC is carried out on the study days, where treatment includes CsA, Tac and placebo respectively in random order. Following an overnight fast the healthy subject / uremic patient arrives in the research laboratory, where a catheter is implanted in each arm for blood sampling and infusion purposes.

Pulse induction: Glucose 6 mg/kg/min is infused every 10 minutes followed by a 9 minute pause. From 30 to 90 min blood is drawn every minute for insulin and every 10th minute for glucose measurements.

First phase insulin secretion: After 120 minutes glucose 0.3 g/kg (maximally 25 g) is infused over 2 min and the catheter is flushed with 50 ml of isotonic saline. Insulin, glucose and c-peptide are measured with a few minutes intervals.

Insulin infusion/HEGC: 1.0 mU/kg/min insulin infusion is initiated at the 165th minute and blood glucose levels are kept at 5.0 mmol/L, using variable infusion of a 20% glucose dilution throughout the following 120 minutes. The final 30 min of the clamp is considered the hyperinsulinaemic steady state period. Aside from glucose, insulin and other endocrinological parameters, measurements of drug concentration and CaN will also be performed.

Perspectives: The studies are expected to give valuable insight into the diabetogenic effects of CI, and to show whether or not CsA and Tac are comparable in their Diabetogenicity. The results will be of relevance to the choice and monitoring of immunosuppressive regimens in kidney transplant recipients as well as the development of better treatment modalities for diabetes.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers (Study 1):

1. Men.
2. Age between 18 years and 50 years. Upper limit can be +2 years if approved by main investigator.
3. Normal OGTT (0 and 120 min test).
4. Body mass index (BMI) 20 - 30 kg/m2. Allowed variations are 5% from the upper and lower limit.
5. Normal serum creatinine and ionisized calcium. Allowed variations are 20% from the upper and lower limit of the normal value for creatinine and 5% for calcium.
6. Normal urine stix
7. Written consent to participate.

Hemodialysis Patients (study 2):

1. Age between 18 years and 70 years. Upper limit can be +2 years if approved by main investigator.
2. BMI < 30 kg/m2. Allowed variations are 5% over the upper limit.
3. On the waiting-list for a kidney transplant.
4. Haemodialysis candidate.
5. Anti-conceptive treatment (contraceptive pill/intrauterine device/patch/ring/ implant/injectable contraceptive) if the patient is a fertile woman.
6. Written consent to participate. -

Exclusion Criteria:

Healthy volunteers (Study 1):

1. Anaemia with haemoglobin levels < 7 mmol/L
2. Participation in any other clinical trial.
3. Subjects who cannot adhere to test conditions.
4. Anamnesis of clinically significant disease, such as:

   * liver disease
   * kidney disease,
   * neurological disease
   * gastrointestinal disease
   * haematological disease
   * endocrine disease
   * lung disease
   * cardiac disease
5. Drug or alcohol abuse, which would render the subject unfit according to the main investigator.
6. Blood donation 1 month prior to the study day
7. Patients with established allergy against CI or other medical products, which might pose a risk if they participated in this study.
8. Use of prescription drugs within one month prior to the study days, unless they are clinically insignificant according to the main investigator.
9. Smoking 8 hours prior to the study day
10. Vigorous exercise 30 minutes prior to the study day.

Hemodialysis Patients (study 2):

1. Peritoneal dialysis.
2. Anaemia with haemoglobin levels < 6 mmol/L.
3. Participation in any other clinical trial.
4. Treatment with corticosteroids, CsA or Tac.
5. Patients who cannot adhere to test conditions.
6. Patients with established allergy against CI or other medical product, which might pose a risk if they participated in this study.
7. Drug or alcohol abuse, which would render the subject unfit according to the main investigator.
8. Anamnesis of current diabetes and/or intake of anti-diabetic medication.
9. Malignancy.
10. Uncontrolled infection.
11. Uncontrolled hypertension.
12. Smoking 8 hours prior to the study day.
13. Vigorous exercise 30 minutes prior to the study day

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | Serial measurements during 120 minute Hyperinsulinemic euglycemic clamp investigation. Performed 3 times on 3 individual days within 4 months after inclusion

SECONDARY OUTCOMES:
insulin secretion | Serial measurements during IVGTT. Performed 3 times on 3 individual days within 4 months after inclusion.
serum free fatty acids | Serial measurements during 5-hour infusions of CsA, Tac or saline. Performed 3 times on 3 individual days within 4 months after inclusion.
serum C-peptide | erial measurements during 5-hour infusions of CsA, Tac or saline. Performed 3 times on 3 individual days within 4 months after inclusion.
blood cyclosporine | erial measurements during 5-hour infusions of CsA, Tac or saline. Performed 3 times on 3 individual days within 4 months after inclusion.
blood tacrolimus | Serial measurements during 5-hour infusions of CsA, Tac or saline. Performed 3 times on 3 individual days within 4 months after inclusion.
respiratory gas exchange, substrate metabolism | Indirect calorimetry performed 3 times on 3 individual days within 4 months after inclusion.
Pulsatile Insulin secretion | erial measurements during glucose entrainment. Performed 3 times on 3 individual days within 4 months after inclusion.
plasma Glucose | erial measurements during 5-hour infusions of CsA, Tac or saline. Performed 3 times on 3 individual days within 4 months after inclusion.
plasma glucagon | erial measurements during 5-hour infusions of CsA, Tac or saline. Performed 3 times on 3 individual days within 4 months after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Aygen Øzbay, MD, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Department of Nephrology, Aarhus University Hospital, Skejby, Aarhus, Jutland, Denmark

REFERENCES:
- [Derived] Ozbay LA, Stubbe J, Jespersen B, Jensen BL. The effects of calcineurin inhibitors on prostanoid synthesis: a randomized cross-over study in healthy humans. Transpl Int. 2013 Feb;26(2):131-7. doi: 10.1111/tri.12004. Epub 2012 Nov 29. PMID 23190385
- [Derived] Ozbay LA, Moller N, Juhl C, Bjerre M, Carstens J, Rungby J, Jorgensen KA. The impact of calcineurin inhibitors on insulin sensitivity and insulin secretion: a randomized crossover trial in uraemic patients. Diabet Med. 2012 Dec;29(12):e440-4. doi: 10.1111/dme.12028. PMID 23003106